CLINICAL TRIAL: NCT05503368
Title: Autologous Cellular Micro-graft in Surgical Treatment of Stable Resistant Vitiligo: A Randomized Self-controlled Trial
Brief Title: Autologous Cellular Graft in Surgical Treatment of Vitiligo
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of availability of the needed kits
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Mogawer, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VS-8822
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Vitiligo, Generalized
Keywords: stable resistant vitiligo; follicular cell suspension; Autologous cellular Micro-grafts; non cultured epidermal suspension
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: self controlled study where 3 comparable lesions will be selected in each patient
Who Masked: Outcomes Assessor
Masking Description: The investigator doing the procedure is the only one who will know which side is assigned to which procedure, but the rest of the investigators including the ones assessing the outcome will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autologous Cellular Micro-grafts suspension added to non cultured epidermal suspension (NCES) (Experimental): Under local anesthesia, a 2.5 mm punch biopsy will be used to extract 3 scalp tissue specimens from the patient's occiput behind the ear, using Rigeneracons medical device (CE certified class I; Human Brain Wave, Turin, Italy). The collected specimens will be placed in Rigeneracons by adding 1.5 mL of sterile physiologic solution to the device. The device then generates a cellular suspension by rotation of Rigeneracons at 80 RPM for 2 minutes. Subsequently, the obtained suspension is diluted with an additional 3 mL sterile physiologic solution. The resulting suspension will be added to NCES and placed on one of the derma braded vitiligo patches
  Interventions: Procedure: surgical treatment of vitiligo using NCES
- Follicle cell suspension added t NCES (Active Comparator): • Under local anesthesia, 1 mm punch will be used to extract hair-follicles from occipital scalp behind the ear. Depending on the area to be transplanted, one hair follicle will be etracted for each 1 cm2. The extracted hair-follicles are washed with phosphate buffered saline (PBS) for about 3 times. The hair-follicles are then incubated with 0.25% trypsin - 0.05% ethylene diamine tetra acetic acid (EDTA) at 37°C for 90 min to prepare the single cell suspension. Within 15-20 min of incubation, the cells start loosening from each other. The hair-follicles are subsequently placed in another tube of trypsin and EDTA. At the end of three such cycles, a thin keratinous shaft is left behind. The cell suspensions of all the tubes are added in a single tube. The final cell pellet is obtained by centrifuging the combined cell suspension at 1000 rpm for 5 min. The resulting suspension will be added to NCES and placed on a comparable derma braded lesion
  Interventions: Procedure: surgical treatment of vitiligo using NCES
- Non cultured epidermal suspension (NCES) (Active Comparator): Melanocyte keratinocyte pellet will be prepared. Donor skin will be harvested from the gluteal region ; using a sterile shaving blade mounted on a Kocher's forceps. Cell Suspension will be prepared by placing the donor skin in 0.25% trypsin-EDTA (GIBCO) solution for 40 minutes at 37 ᴼC. sample and trypsin will be poured into a labelled petri dishes then neutralized using ringer's lactate. All the steps will be performed in a laminar air flow bench under strict aseptic conditions. The epidermis will be detached from the dermis which will be discarded. Then the epidermis will be cut into tiny pieces and scrapped so that no pigment is left on the surface. Afterwards, they will be transferred to sterile falcon tubes and centrifuged for 10 minutes at 1,000 rpm. The floating epidermal fragments and supernatant fluid will be removed, leaving the cell pellet containing epidermal cells rich in melanocytes and Keratinocytes at the bottom.
  Interventions: Procedure: surgical treatment of vitiligo using NCES

INTERVENTIONS:
Procedure: surgical treatment of vitiligo using NCES — NCES is the standard technique for surgical treatment of vitiligo, herein we compare the standard technique, to added autologous cellular micro-grafts and to follicle cell suspension

SUMMARY:
This is a double blinded self controlled randomized trial to assess Autologous Micro Cellular Grafts in surgical treatment of stable resistant vitiligo. Given the stem cells, progenitor cells, and growth factors rich hair follicle based suspension resulting from Autologous Cellular Micro grafts (ACM), we aim at assessing the efficacy of ACM generated suspension in comparison to follicle cell suspension in surgical treatment of stable resistant vitiligo.

DETAILED DESCRIPTION:
Prior to surgery, two comparable lesions will be selected.

Lesions will be assessed for:

1. Surface Area using point counting technique.
2. Any attempts of pigmentation using VESTA score. Lesions will be derma braded under local anesthesia using fractional laser CO2 resurfacing, Using dot mode off resurfacing will be performed at a power of 18-20 W, dwell time 1,000 milliseconds (DEKA, Florence, Italy). One to three passes will be performed until the epidermis is removed uniformly.

Autologous Cellular Micrografts (ACM) suspension generated by regenera technique Under local anesthesia, a 2.5 mm punch biopsy will be used to extract 3 scalp tissue specimens from the patient's occiput behind the ear, using Rigeneracons medical device (CE certified class I; Human Brain Wave, Turin, Italy). The collected specimens will be placed in Rigeneracons by adding 1.5 mL of sterile physiologic solution to the device. The device then generates a cellular suspension by rotation of Rigeneracons at 80 RPM for 2 minutes. Subsequently, the obtained suspension is diluted with an additional 3 mL sterile physiologic solution. The resulting suspension will be added to melanocyte pellet generated by NCES technique and will be spread on one of the derma braded vitiliginous patches.

Non cultured Epidermal Suspension (NCES):

Melanocyte keratinocyte pellet will be prepared. Donor skin will be harvested from the gluteal region after anaesthetizing the area with intra-lesional Mepicaine L; using a sterile shaving blade mounted on a Kocher's forceps. An expansion ratio of 1:2 was used for each lesion separately to ensure equivalent melanocyte concentration in all transplanted lesions. Cell Suspension will be prepared by placing the donor skin in 0.25% trypsin-EDTA (GIBCO) solution for 40 minutes at 37 ᴼC. Each sample and trypsin will be poured into a labelled petri dishes then neutralized using ringer's lactate. All the steps will be performed in a laminar air flow bench under strict aseptic conditions. The epidermis will be detached from the dermis which will be discarded. Then the epidermis will be cut into tiny pieces and scrapped so that no pigment is left on the surface. Afterwards, they will be transferred to two labelled sterile falcon tubes and centrifuged for 10 minutes at 1,000 rpm. The floating epidermal fragments and supernatant fluid will be removed, leaving the cell pellet containing epidermal cells rich in melanocytes and Keratinocytes at the bottom. The resultant pellet will be suspended once in ACM generated by regenera technique, once in hair follicle suspension and once in 1 ml of ringer's lactate.

Follicular Cellular Suspension:

* Under local anesthesia, 1 mm punch will be used to extract hair-follicles from occipital scalp behind the ear. Depending on the area to be transplanted, one pigmented follicles will be extracted for each 1 cm2. The extracted hair-follicles are washed with phosphate buffered saline (PBS) for about 3 times. The hair-follicles are then incubated with 0.25% trypsin - 0.05% ethylene diamine tetra acetic acid (EDTA) at 37°C for 60 min divided in to 3 intervals to prepare the single cell suspension. The first interval lasted 30 minutes after which the supernatant fluid containing separated cells was poured into a new falcon tube and neutralized by 1% fetal bovine serum. Fresh trypsin was then added to hair follicles and reincubated for 15 minutes twice.
* At the end of three such cycles, a thin keratinous shaft is left behind. The cell suspensions of all the tubes are added in a single tube. The final cell pellet is obtained by centrifuging the combined cell suspension at 1000 rpm for 5 min. The resulting suspension will be added to melanocyte pellet generated by NCES technique and will be spread on a comparable derma braded lesion.

The resultant suspension will be checked for melanocyte count and viability using trypan blue dye exclusion method to ensure above 250 viable cells/mm2 of the recipient area prior to its spreading on the derma braded vitiligo patch.

Both sites will be covered with a dry collagen sheet followed by sterile surgical pad and tegaderm.

The area will be immobilized after bandaging and the patient will be advised to restrict movement at the operated site.

Patients will start a 1-week course of antibiotics. Dressings will be removed after 1 week, and patients will receive excimer laser sessions, 3 sessions per week for 3 months.

Patients will be followed up monthly for 3 months following the first visit at 1 week.

At 3 months, both qualitative and quantitative assessment will be done. Qualitatively, blinded physician assessment of repigmentation as well as color match using serial photographs will be done. Quantitatively, point counting method as well as VESTA score will be used as well to assess degree of repigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-segmental vitiligo (NSV) / segmental resistant lesions; with either 2 comparable lesions or large patches that can be divided
* Stability for ≥ 1 year
* Age >18 years
* Lack of treatment for at least 1 month prior to surgery.

Exclusion Criteria:

* -Vitiligo lesions responsive to conventional treatment modalities
* Active vitiligo; new lesions, expansion of old lesions or koebnerization in < 1 year
* Age < 18 years.
* Keloidal tendency
* Bleeding tendency
* Pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
comparing change in surface area in three arms | 3 months follow up are required to assess response
  Percent change in surface area calculated by point counting technique will be compared between three arms

SECONDARY OUTCOMES:
comparing percent of repigmentation in three arms | 3 months follow up are required to assess response
  Percent change in lesional pigmentation as per VESTA score will be compared between three arms

CONTACTS AND LOCATIONS:
Overall Officials: Rania M Mogawer, Principal Investigator — Kasr Alainy, Cairo University Hospitals; Samia M Esmat, Study Director — Kasr Alainy, Cairo University Hospitals
Locations (1):
- Cairo university hospitals, dermatology outpatient clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Participants' data that underlie reported results will be shared upon request, after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 12 months after article publication
Access Criteria: Controlled Access:
  Researchers who provide a methodologically sound proposal will be allowed to access data to achieve aims in the approved proposal.

REFERENCES:
- [Result] El-Zawahry BM, Esmat S, Bassiouny D, Zaki NS, Sobhi R, Saleh MA, Abdel-Halim D, Hegazy R, Gawdat H, Samir N, El-Hawary M, El Maadawi Z, Gouda H, Khorshied M. Effect of Procedural-Related Variables on Melanocyte-Keratinocyte Suspension Transplantation in Nonsegmental Stable Vitiligo: A Clinical and Immunocytochemical Study. Dermatol Surg. 2017 Feb;43(2):226-235. doi: 10.1097/DSS.0000000000000962. PMID 28157763
- [Result] Ruiz RG, Rosell JMC, Ceccarelli G, De Sio C, De Angelis GC, Pinto H, Astarita C, Graziano A. Progenitor-cell-enriched micrografts as a novel option for the management of androgenetic alopecia. J Cell Physiol. 2020 May;235(5):4587-4593. doi: 10.1002/jcp.29335. Epub 2019 Oct 23. PMID 31643084
- [Result] Zari S. Short-Term Efficacy of Autologous Cellular Micrografts in Male and Female Androgenetic Alopecia: A Retrospective Cohort Study. Clin Cosmet Investig Dermatol. 2021 Nov 19;14:1725-1736. doi: 10.2147/CCID.S334807. eCollection 2021. PMID 34824538
- [Result] Razmi T M, Kumar R, Rani S, Kumaran SM, Tanwar S, Parsad D. Combination of Follicular and Epidermal Cell Suspension as a Novel Surgical Approach in Difficult-to-Treat Vitiligo: A Randomized Clinical Trial. JAMA Dermatol. 2018 Mar 1;154(3):301-308. doi: 10.1001/jamadermatol.2017.5795. PMID 29387874
- [Result] Thakur V, Kumar S, Kumaran MS, Kaushik H, Srivastava N, Parsad D. Efficacy of Transplantation of Combination of Noncultured Dermal and Epidermal Cell Suspension vs Epidermal Cell Suspension Alone in Vitiligo: A Randomized Clinical Trial. JAMA Dermatol. 2019 Feb 1;155(2):204-210. doi: 10.1001/jamadermatol.2018.4919. PMID 30601885
- [Result] Mohanty S, Kumar A, Dhawan J, Sreenivas V, Gupta S. Noncultured extracted hair follicle outer root sheath cell suspension for transplantation in vitiligo. Br J Dermatol. 2011 Jun;164(6):1241-6. doi: 10.1111/j.1365-2133.2011.10234.x. PMID 21275943
- [Result] Gho CG, Braun JE, Tilli CM, Neumann HA, Ramaekers FC. Human follicular stem cells: their presence in plucked hair and follicular cell culture. Br J Dermatol. 2004 May;150(5):860-8. doi: 10.1111/j.1365-2133.2004.05862.x. PMID 15149497